CLINICAL TRIAL: NCT06409195
Title: Open-Label Study of the Safety and Efficacy of SM-020 Gel 1.0% in Subjects With Seborrheic Keratoses and Non-Melanoma Skin Cancers (Basal Cell Carcinoma and Squamous Cell Carcinoma In Situ)
Brief Title: A Trial to Study the Safety and Efficacy of SM-020 Gel 1.0% in Subjects With Seborrheic Keratoses and Non-Melanoma Skin Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: DermBiont, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT-217
Record Dates: First submitted 2024-04-15; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Non-Melanoma Skin Cancers
MeSH Terms: interventions — Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Cohort 1: SM-020 gel 1.0% BID for 28 days to superficial BCCs
  Interventions: Drug: SM-020 1% Gel
- Cohort 2 (Experimental): Cohort 2: SM-020 gel 1.0% BID for 28 days to nodular BCCs
  Interventions: Drug: SM-020 1% Gel
- Cohort 3 (Experimental): Cohort 3: SM-020 gel 1.0% BID for 28 days to infiltrating BCCs
  Interventions: Drug: SM-020 1% Gel
- Cohort 4 (Experimental): Cohort 4: SM-020 gel 1.0% BID for 28 days to SCCISs
  Interventions: Drug: SM-020 1% Gel
- Cohort 5 (Experimental): Cohort 5: SM-020 gel 1.0% BID for 28 days to SKs
  Interventions: Drug: SM-020 1% Gel

INTERVENTIONS:
Drug: SM-020 1% Gel — SM-020 gel 1.0% will be applied topically. Subjects will be treated with twice daily application to at least 1 and up to 5 Target Lesions (TLs) for 28 days.

SUMMARY:
Open-Label study evaluating safety and efficacy of SM-020 Gel 1.0% in subjects with Seborrheic Keratoses and Non-Melanoma Skin Cancers (i.e. Basal Cell Carcinoma and Squamous Cell Carcinoma In Situ). Subjects will be enrolled into 1 of 5 cohorts. Each cohort will enroll approximately 5-10 subjects with at least 1 eligible lesion to be treated. A maximum of 5 lesions may be enrolled per subject. Treatment for all subjects and all lesions will be twice daily for approximately 28 days. Post treatment, residual lesions may be excised per standard of care for histological evaluation. The duration of the study is estimated to be approximately up to 12 weeks from the beginning of the Screening period until the last subject's last visit.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study:

1. Must be able to comprehend and willing to sign an informed consent form (ICF).
2. Must complete a signed Health Information Portability and Accountability Act (HIPAA) authorization form which permits the use and disclosure of the subject's individually identifiable health information.
3. Must be at least 18 years of age.
4. Histologically confirmed seborrheic keratosis, basal cell skin cancer (superficial, nodular, and/or infiltrating subtype) and/or squamous cell carcinoma in situ from screening biopsies
5. At least 1 and up to 5 screened and histologically confirmed eligible NMSC and/or SK lesions max between 0.5-2.0 cm in greatest tumor diameter
6. NMSCs must also meet the following criteria:

   Primary tumor (no recurrent or previously treated tumors)

   Located on the scalp, face (excluding ears and nose), trunk, or extremities (excluding the hands and feet)

   Qualifies for standard surgical excision or Mohs micrographic surgery as primary therapy

   Not be on the eyelid or within 5 mm of the orbital rim
7. SKs must also meet the following criteria

   PLA 2 (<1 mm in thickness)

   Have one or more of the following dermoscopy features throughout the entirety of the lesion: crypts (comedo-like openings), milia cysts, hairpin vessels with white halo, fat sharp demarcation, blue-white pigmentation/veil as long as milia and crypts are present within, more than one color, cerebriform structure (gyri and sulci/network-like pattern/ridges and fissures/fat fingers), irregular vessels (inframammary only), granularity at periphery, stalactite/Tsingy pattern, plate-like/fractured pattern (Simionescu et al., 2012) (Note: SK lesions must NOT have any of the following features indicative of malignancy under dermoscopy: pinpoint vessels, smooth blue-white pigmentation/veil without milia or crypts within, hairpin vessels without white halo, white artifacts, irregular vessels (except for inframammary lesions). Additionally, SK lesions must not have a moth-eaten border or fingerprint structures indicative of lentigos or a network pattern indicative of a melanocytic lesion)

   Located on the scalp, face (including ears), trunk, intertriginous areas, or extremities

   Not be on the eyelid or within 5 mm of the orbital rim
8. Must be free of any known disease state or physical condition which, in the Investigator's opinion, might impair evaluation of any treated lesion or which exposes the subject to an unacceptable risk by study participation.
9. Must be willing and able to follow all study instructions and to attend all study visits.
10. Technical ability to apply treatment to all enrolled lesion
11. Must be willing to have all lesions removed surgically by either Mohs micrographic surgery or standard excision for NMSCs or shave excision for SKs at the final 2-week follow up visit.

Exclusion Criteria:

Subjects meeting any of the following criterion will be ineligible and excluded from this study:

1. Positive urine pregnancy test, pregnant, lactating, or female of childbearing potential who does not agree to use an active method of birth control (such as oral contraceptive pills (OCPs), Intrauterine devices (IUDs), birth control implants, vaginal rings, or injections) for the duration of the study.
2. SK lesions that are clinically atypical and/or rapidly growing in size or number.
3. Presence of multiple eruptive SK lesions (sign of Leser-Trelat)
4. Current systemic malignancy.
5. Past history of lymphoproliferative disorder
6. Any use of the following systemic therapies within the specified period prior to the Baseline visit and while on study:

   Retinoids; 180 days

   Chemotherapy; 180 days

   Immunosuppressive therapy; 28 days

   Biologics (e.g., interferon, interferon inducers, or immunomodulators such as such as Tumor necrosis factor (TNF) inhibitors; Interleukin (IL) inhibitors; B-cells inhibitors; and T-cells inhibitors and other immunomodulatory systemic biologics such as Anti-TNF biologics including: adalimumab (Humira®), certolizumab pegol (Cimzia®), etanercept (Enbrel®), golimumab (Simponi®) and infliximab (Remicade®), and Non-TNF biologics including: abatacept (Orencia®), anakinra (Kineret®), rituximab (Rituxan®), tolcilizumab (Actemra®), tofacitinib (Xeljanz®), and ustekinumab (Stelara®)); 28 days

   Glucocorticosteroids (Oral and intramuscular); 28 days

   Anti-metabolites (e.g., methotrexate); 28 days

   Vismodegib; 180 days

   Subjects taking known photosensitizing medications or CYP3A inhibitors (see Section 6.10 for more details); 28 days
7. Any use of the following topical therapies within the specified period prior to the Baseline visit and while on study on or in a close proximity to any treated lesion (TL) that, in the Investigator's opinion, could interfere with the investigational product study treatment applications or the study assessments:

   Laser, light or other energy-based therapy [e.g., intense pulsed light (IPL), photo-dynamic therapy (PDT)]; 180 days

   Liquid nitrogen, electrodessication, curettage, imiquimod, 5-fluorouracil, or ingenol mebutate; 180 days

   Retinoids; 28 days

   Microdermabrasion or superficial chemical peels; 28 days

   Glucocorticosteroids or antibiotics; 28 days
8. Occurrence or presence of any of the following within the specified period prior to the Baseline visit on or in the proximity of any TL that, in the Investigator's opinion, could interfere with the investigational product study treatment applications or the study assessments:

   Cutaneous malignancy: 180 days (excluding those to be enrolled)

   Sunburn; currently

   Body art (e.g., tattoos, piercing, etc.); currently
9. History of sensitivity to any of the ingredients in the investigational product.
10. Any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or other condition(s) (e.g., sunburn, excessive hair, open wounds, lupus, photosensitive disorders etc.) that, in the opinion of the Investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations.
11. Participation in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to the Screening visit.
12. History of hypertrophic scarring or keloid formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of lesions that achieve a 50% reduction in greatest diameter of cohort-assigned TL(s) at week 6 compared to baseline | At week 6
Safety and Tolerability will be evaluated through assessment of the severity of the signs and symptoms of Application Site Reactions (ASRs) | Screening, Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, and Week 8
  Application Site Reactions will be evaluated based on the severity of the signs and symptoms of pain, burning, stinging, pruritus, erythema, edema, exudation, erosion/ulceration, hyperpigmentation,and hypopigmentation.
Safety and Tolerability as evaluated by review of adverse events | Screening, Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, and Week 8
  Grade 1 = Mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated Grade 2 = Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL Grade 3 = Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL Grade 4 = Life-threatening consequences: urgent intervention indicated Grade 5 = Death related to AE with Grade 1 being the minimum value and Grade 5 being the maximum value, with a higher value indicating higher severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology, Laser and Vein Specialist, Charlotte, North Carolina, United States